CLINICAL TRIAL: NCT00172458
Title: Clinical Results and Restenosis Analysis of Symptomatic Ostial Vertebral Artery Stenosis Treated With Tubular Coronary Stents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700454
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-08

CONDITIONS: Vertebral Artery Stenosis
MeSH Terms: conditions — Vertebrobasilar Insufficiency

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Vertebral artery stenosis (VAS) decreases posterior brain perfusion, causing vertebrobasilar insufficiency (VBI). It is also an important embolic source to the posterior brain. The most frequently involved location is the proximal part of the vessel, including the ostium. Various surgical procedures have been described for the treatment of proximal VAS with symptoms refractory to medical therapy, but all are technically difficult with high operative mortality and morbidity.

Endovascular intervention has been described as an alternative to surgery. Balloon angioplasty is limited by elastic recoil and dissection. The restenosis rates reported in the literature varied, as high as 75 %. Stenting offers salvage following unsuccessful balloon angioplasty, and primary stenting have been shown to be safe and effective with lower restenosis rate. Coronary equipments are ideal for ostial VAS, considering the size of the artery and location of the lesion. Recently, Albuquerque et al. reports a relative high restenosis rate in a longer follow-up duration. Restenosis seems to become an important issue regarding the patients' quality of life. However, there is no clinical parameter to predict restenosis of VAS. The purpose of this study is to evaluate the clinical results of our series of symptomatic ostial VAS treated exclusively with tubular balloon expandable coronary stents. We sought to identify predictors of restenosis.

This is a clinical observation study. Only chart review and angiographic review will be performed.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic vertebral artery stenosis treated by stenting

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Hesien-Li Kao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan